CLINICAL TRIAL: NCT07225062
Title: Improving HIV Prevention and Substance Use Post-Sexual Assault Services for Adolescents and Young Adults
Brief Title: Improving HIV Prevention and Substance Use Post-Sexual Assault Services
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Diane Santa Maria, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSC-SN-25-0423
Record Dates: First submitted 2025-11-03; First posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: HIV Infections; Substance Use; Sexual Assault
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data collectors will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced intervention (Experimental)
  Interventions: Behavioral: Enhanced intervention
- Usual Care (Active Comparator)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Enhanced intervention — The intervention has three components: 1). Exploring how to increase access to and promotion of SANE services among vulnerable AYA within the 72 hr window for nPEP treatment; 2). Enhanced SANE services to increase same-day access to nPEP and DoxyPEP and 3). An advocate-delivered screening, brief intervention, and referral to prevent and address substance misuse.
  Arms: Enhanced intervention
Behavioral: Usual Care — The usual care condition will be used with control participants and entail receiving typical SANE services without modifications to enhance HIV prevention or substance use screening, brief intervention, or referral to treatment
  Arms: Usual Care

SUMMARY:
The purpose of this study is to tailor existing sexual assault nurse examiner (SANE) services with same-day HIV prophylaxis and substance use screening, brief intervention, or referral using semi-structured adolescents and young adults (AYA) survivor and key informant interviews, and iterative co-design/pilot testing of adapted strategies with the youth working group (YWG), to optimize study mechanisms and outcome measures using cognitive interviews, analysis of community partner data, and recruitment and retention strategies with the youth working group (YWG) and community advisory board (CAB), to conduct a pilot randomized controlled trial with 40 AYA to test feasibility, acceptability, and initial efficacy compared to usual care, to evaluate recruitment, randomization, and follow-up strategies; adherence to intervention dose; retention benchmarks; and acceptability and to evaluate preliminary efficacy of outcome measures (uptake of post-assault HIV prevention and substance use treatment).

ELIGIBILITY:
Inclusion Criteria:

* experienced a sexual assault within the last 72 hours
* speak English
* not planning to move out of the metro area during the study.

Exclusion Criteria:

* noticeably intoxicated or under the influence
* are overtly having severe, untreated mental illness symptoms

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2027-01-04 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment feasibility as measured by percentage of eligible individuals screened | end of study (1 month after baseline)
Recruitment feasibility as measured by percentage of eligible individuals enrolled | end of study (1 month after baseline)
Recruitment feasibility as measured by time delay from screening to enrollment | end of study (1 month after baseline)
Recruitment feasibility as measured by time to enroll sufficient sample size | end of study (1 month after baseline)
Recruitment feasibility as measured by percentage loss to exclusion criteria. | end of study (1 month after baseline)
Randomization strategies as measured by proportion randomized to intervention and control | end of study (1 month after baseline)
Retention as measured by the number of participants that completed the one month follow-up survey | end of study (1 month after baseline)
Retention of the intervention group as measured by the number of participants that completed the one month follow-up survey | end of study (1 month after baseline)
Retention of the control group as measured by the number of participants that completed the one month follow-up survey | end of study (1 month after baseline)
Adherence to intervention as measured by percentage of content completed in the fidelity checklist | end of study (1 month after baseline)
Acceptability as measured by percentage of data loss | end of study (1 month after baseline)
Acceptability as measured by score on the credibility/expectancy questionnaire | end of study (1 month after baseline)
  The Credibility and Expectancy Questionnaire (CEQ) was used to assess the acceptability of the intervention. All participants completed both subscales: the credibility subscale and the expectancy subscale. Each subscale total score ranges from 0 to 10, with higher scores indicating greater perceived acceptability. The expectancy subscale is reported.
Acceptability as measured by score on the credibility/expectancy questionnaire | end of study (1 month after baseline)
  The Credibility and Expectancy Questionnaire (CEQ) was used to assess the acceptability of the intervention. All participants completed both subscales: the credibility subscale and the expectancy subscale. Each subscale total score ranges from 0 to 10, with higher scores indicating greater perceived acceptability. The credibility subscale is reported.

SECONDARY OUTCOMES:
Uptake of post-assault HIV prevention as measured by self report of nPEP uptake | 1-month follow-up
Uptake of substance use treatment as self reported as reported on the self report questionnaire | 1-month follow-up
Uptake of post-assault HIV prevention as measured by self report of Doxycycline Post-Exposure Prophylaxis (DoxyPEP) uptake | 1-month follow-up
Adherence of non-occupational Post-Exposure Prophylaxis (nPEP) as reported on the self report questionnaire | 1-month follow-up
Adherence of substance use treatment as reported on the self report questionnaire | 1-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Diane M Santa Maria, DrPH,MSN,FAANRN,PHNA-BC,FSAHM, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No